CLINICAL TRIAL: NCT00684242
Title: A Pilot Clinical Trial of Lenalidomide (Revlimid®) for the Treatment of Refractory Cancer Pain
Brief Title: Lenalidomide (Revlimid) for the Treatment of Refractory Cancer Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0750
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2012-12

CONDITIONS: Advanced Cancer; Pain
Keywords: Advanced Cancer; Refractory Cancer Pain; Lenalidomide; Revlimid; CC-5103
MeSH Terms: conditions — Pain; Cancer Pain | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide (Experimental): 10 mg by mouth daily
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 10 mg by mouth daily
  Other Names: Revlimid; CC-5103

SUMMARY:
The goal of this clinical research study is to learn if lenalidomide can help to treat uncontrolled pain caused by advanced cancer.

Primary Objectives:

1. Determine efficacy of Lenalidomide for the treatment of refractory cancer pain, as measured by the change on Edmonton symptom assessment scale (ESAS).

Secondary Objectives:

1. To determine the effect of Lenalidomide on fatigue, sleep, depressed mood, nausea and appetite/anorexia.
2. Determine changes in serum levels of inflammatory cytokines (IL-1beta, IL-6, TNF-alpha, interferon(IFN)-alpha and IFN-gamma, and C-reactive protein) before and after treatment with Lenalidomide.
3. Effect of Lenalidomide on T-cell subsets especially T-regulatory cells
4. Effect of Lenalidomide on the expression of costimulatory receptors, CD80, CD86, and CD40, on myeloid and plasmacytoid dendritic cells
5. Safety (type, frequency, severity, and relationship of adverse events to study treatment)

DETAILED DESCRIPTION:
The Study Drug:

Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells. The drug is also designed to decrease the level of certain proteins in the blood called cytokines, which may result in decreased pain.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take lenalidomide capsules each morning, with or without food. Take lenalidomide capsules whole, with a 4-ounce (1/2 cup) glass of water at the same time each day. Do not break, chew, or open the capsules. If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose).

If you take too much lenalidomide, call your study doctor or health care provider or poison control center right away.

You will also be allowed to take strong pain killers such as morphine as prescribed by your study doctor for pain. If you need more than 3 doses of these pain killers in a 24-hour period, you should call your study doctor.

Study Visits:

You will visit the clinic throughout the study. At each visit, you will be asked to return any unused study drug and empty bottles to the clinic and you will be asked about any side effects you may be experiencing. The last study visit will be on Day 43 or Day 57, depending on the side effects you may experience. The following tests and procedures will be performed:

On Day 8:

Blood (about 1 tablespoon) will be drawn for routine tests and women who are able to have children will have a blood pregnancy test.

Day 15:

Blood (about 1 tablespoon) will be drawn for routine tests. Women who are able to have children will have a blood (1-2 teaspoons) pregnancy test. You will complete 5 questionnaires about the pain, the pain symptoms, and any side effects you may be having. The questionnaires will take about 30 to 40 minutes to complete. Women who are able to have children will have a blood pregnancy test.

Day 22:

Blood (about 1 tablespoon) will be drawn for routine tests. Women who are able to have children will have a blood (1-2 teaspoons) pregnancy test.

Day 29:

You will complete the same questionnaires as on Day 15. Women who are able to have children will have a blood pregnancy test and will be counseled about pregnancy precautions and risks. Blood (about 1 tablespoon) will be drawn for routine tests. Women who are able to have children will have a blood (1-2 teaspoons) pregnancy test.

Day 36:

Blood (about 1 tablespoon) will be drawn for routine tests.

Day 43:

Blood (about 1 tablespoon) will be drawn for routine tests. You will complete the same questionnaires as on Day 15. If this is your last visit, you will have an ECG. Women who are able to have children will have a blood (1-2 teaspoons) pregnancy test.

Day 57 (if necessary):

You will complete the same questionnaires as on Day 15. Blood (about 1 tablespoon) will be drawn for routine tests. You will complete the same questionnaires as on Day 15. If this is your last visit, you will have an ECG. Women who are able to have children will have a blood (1-2 teaspoons) pregnancy test.

Day 71 (if necessary):

If you stopped taking the drug on Day 57, a blood (1-2 teaspoons) pregnancy test will be done.

Length of Study:

You may take lenalidomide for up to 57 days. You will be taken off study if the disease gets worse or if intolerable side effects occur.

If you are a female who is able to have children and you do take lenalidomide for all 57 days, you will be required to have a blood (1-2 teaspoons) pregnancy test 28 days after your last dose of lenalidomide.

The routine blood draws on Days 8, 22, and 36 may done at your home (by a study nurse), local doctor's office, or at M. D. Anderson.

All patients who were on lenalidomide and then stopped taking it, will be checked every 3 to 5 weeks for a period of 1 year. During the follow-up visits, certain tests and procedures will be performed. These include a symptom questionnaire, blood draw for routine tests, a check of your side effects, and pregnancy testing for women who are still able to become pregnant. These are the same tests that were done while you were on the study.

Daily Drug Diary and Questionnaire:

Starting on Day 1 until the end of the study, you will complete a questionnaire once daily about any symptoms and pain you may be experiencing. It will take about 5 minutes to complete each time. You will also be provided with a drug diary to write down when and how often you take pain medication. You should bring your completed diary to each study visit so it can be reviewed by the research nurse.

Phone Call Follow-up:

You will be contacted by telephone at home to be asked questions about your symptoms and any side effects you may have experienced. You will be called on Day 8 (plus or minus 3 days), Day 22 (plus or minus 3 days) and Day 36 (plus or minus 3 days). The phone calls will last about 10-15 minutes each time.

End-of-Study Visit:

You will come to the clinic 28 days after your last dose of lenalidomide for a follow-up visit. You will be checked for side effects, and women who are able to have children must have a negative blood (1-2 teaspoons) pregnancy test.

This is an investigational study. Lenalidomide is approved by FDA for the treatment of myelodysplastic syndrome (MDS) and in combination with dexamethasone for patients with multiple myeloma (MM). Lenalidomide is not FDA approved for pain relief. Its use in this study is investigational. If you experience intolerable pain after you stop receiving the study drug, you will be allowed to start receiving lenalidomide (off study). You will be monitored for side effects for every 2-3 weeks while you are on this medication for a period of 1 year. Up to 15 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer with a diagnosis of refractory cancer pain (Refractory cancer pain is defined for research purposes as the pain secondary to cancer that is refractory to strong opioids as determined by the persistence of pain despite at least 2 or more opioid escalation and/ or opioid rotations for a given pain syndrome).
2. Pain intensity score of 5 or greater on Edmonton Symptom Assessment scale.
3. Understand and voluntarily sign an informed consent form.
4. Age >/=18 years at the time of signing the informed consent form.
5. Able to adhere to the study visit schedule and other protocol requirements.
6. Patients who are receiving chemotherapy are eligible for study if approved by primary oncologist. The PI or enrolling physician will obtain and document approval from the primary oncologist in the patient's study documents.
7. Will consent to the use of asprin (81 or 325 mg) or Low molecular weight heparin (if intolerant to to asprin)
8. Laboratory test results within these ranges within the past 14 days: Absolute neutrophil count >/= 1.5 * 10^9/L , Platelet count >/= 100 * 10^9/L, Serum creatinine </= 2.0 mg/dL, Total bilirubin </=1.5 mg/dL, and aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) </=2 * Upper limit of normal (ULN) or </= 5 * ULN if hepatic metastases are present.
9. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
10. Females of childbearing potential (FCBP). A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
11. FCBP must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 to 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide.
12. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix : Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. A history of development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concomitant use of sargramostim (GM-CSF), including radiation, thalidomide, or other investigational agents is not permitted while subjects are receiving study drug during the treatment portion of the study.
9. Known positive for HIV or infectious hepatitis, type A, B or C.
10. Patients with known myeloid malignancy or tumors having bone marrow involvement.
11. History of alcohol abuse as determined by the CAGE questionnaire (> / = 2/4).
12. Individual with clinically evident impaired cognition.
13. Patient with a history of psychiatric diagnosis of depression or clinical diagnosis of depression as determined by the treating physician or Hospital Anxiety Depression Scale total score of 13 or greater.
14. All major surgeries such as thoracotomy etc., that requires wound healing within last 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennurajalingam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 22, 2008 to November 1, 2010. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: One participant was enrolled but excluded from the trial before assignment to groups.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 3
Age Continuous [Median (Full Range); unit: years] | 64 [44 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Cancer Pain Intensity Determined by Edmonton Symptom Assessment Scale (ESAS)
Description: Changes in cancer pain from baseline to day 15 using ESAS to measure participant responses to 10 common symptoms (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, appetite, sleep problems, and feeling of well-being). Intensity of symptoms rated on a 0 to 10 scale from 0 "no symptom" to 10 "worst possible symptom."
Time Frame: From baseline to Day 15
Population: One participant was not evaluable for Day 15.
Measure: Number; unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
units on a scale
  Participant 1 | 0
  Participant 2 | -2

ADVERSE EVENTS:
Time Frame: 1 year and 8 months
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=3)
Constipation (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (Extremity-Limb) (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=3)
Constipation (Gastrointestinal disorders) | 2 (6)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dry Mouth (General disorders) | 2 (3)
Fatigue (General disorders) | 3 (9)
Insomnia (General disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (8)
Pain (Extremity-Limb) (Gastrointestinal disorders) | 1 (1)
Pain (NOS) (General disorders) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 (2)
Somnolence (General disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (2)
Watery Eye (Eye disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No